CLINICAL TRIAL: NCT03544905
Title: A Multi-center, Open-label, Single Arm, Dose Escalation and Dose Extension Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of CYH33 in Advanced Solid Tumors Patients.
Brief Title: Study to Evaluate the Safety, Tolerate, Pharmacokinetics and Preliminary Efficacy of CYH33
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Haihe Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CYH33-101
Record Dates: First submitted 2018-05-22; First posted 2018-06-04 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — CYH33; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dose escalation study of CYH33 (Experimental): To determine the maximum tolerated dose (MTD) of CYH33
  Interventions: Drug: CYH33 for tablet

INTERVENTIONS:
Drug: CYH33 for tablet — 1mg; 5mg; 10mg; 20mg; 30mg; 50mg; 75mg; 100mg; 130mg; 160mg; 200mg; 240mgBID or QD(Decided by SMC accroding to the safty and PK data)

SUMMARY:
This study is a Multi-center, Open-label, single arm, Dose Escalation and Dose Extension Phase 1 Study to Evaluate the Safety , Tolerability, Pharmacokinetics and Preliminary Efficacy of CYH33 in Advanced Solid Tumors Patients.

DETAILED DESCRIPTION:
This study includes Phase Ia and Phase Ib.

In the dose climbing part of phase Ia, the safety, tolerance and pharmacokinetics characteristics of CYH33 in patients with advanced solid tumors who failed to receive standard treatment, did not tolerate or did not have standard treatment at present will be observed to determine MTD; Before determining MTD, select safe and highly reliable and effective dose levels for simultaneous expansion. Phase Ia dose expansion includes patients with advanced solid tumors who have failed to undergo standard treatment, who are intolerant of PIK3CA gene mutation, or who do not have standard treatment at present, to further evaluate safety, tolerance and initial efficacy.

In Phase Ib, the safety and preliminary efficacy of CYH33 on patients with advanced breast cancer, ovarian cancer, endometrial cancer, cervical cancer, head and neck squamous cell carcinoma, esophageal and gastroesophageal junction squamous cell carcinoma, ovarian clear cell carcinoma and other solid tumors with PIK3CA gene mutation who have failed, are intolerant or do not have standard treatment at present will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* main inclusion:

  1. Evidence of a personally signed informed consent document;
  2. Male and/or female subjects above the ages of 18 years;
  3. Locally advanced or metastatic solid tumor patients who have failed or relapsed on current standard of care for Phase 1a;
  4. Subject may provide Tumor tissue section(at least 8 pieces) if they agree;
  5. ECOG performance score 0-1;
  6. Life expectancy ≥ 12 weeks;
  7. At least 1 measurable target lesion on the baseline scan as per RECIST 1.1

Exclusion Criteria:

* main criteria:

  1. prior received anti-tumor treatment, including anticancer drugs for the treatment within 28 days of first dose of study treatment;
  2. Prior or concomitant other malignant tumor;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2018-07-05 (Actual); Primary Completion 2024-12-04 (Actual); Study Completion 2024-12-04 (Actual)

PRIMARY OUTCOMES:
MTD(Max tolerance does) | 35 days
  To evaluate the MTD in patients with advanced solid tumor

CONTACTS AND LOCATIONS:
Overall Officials: Ruihua Xu, M.D, Principal Investigator — Sun Yat-sen University
Locations (30):
- China (30):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Lu'an People's Hospital, Lu'an, Anhui
  - Lu'an Hospital of Traditional Chinese Medicine, Lu'an, Anhui
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Chongqing Cancer Hospital, Chongqing, Chongqing Municipality
  - Xiang'an Hospital of Xiamen University, Xiamen, Fujian
  - Dongguan People's Hospital, Dongguan, Guangdong
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Yuebei People's Hospital, Shaoguan, Guangdong
  - Shenzhen Hospital of Cancer Hospital, Chinese Academy of Medical Sciences, Shenzhen, Guangdong
  - Liuzhou Workers Hospital, Liuchow, Guangxi
  - Affiliated Tumor Hospital of Guangxi Medical University, Nanning, Guangxi
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Anyang Cancer Hospital, Anyang, Henan
  - Nanyang First People's Hospital, Nanyang, Henan
  - The First Affiliated Hospital of Nanyang Medical College, Nanyang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Hunan Province Directly Affiliated Traditional Chinese Medicine Hospital, Zhuzhou, Hunan
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Obstetrics and Gynecology Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Dali University, Dali, Yunnan
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang